CLINICAL TRIAL: NCT02365753
Title: Effect of Pulsed Electromagnetic Field Therapy on Pain After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Donald Phillibert, Attending Phyisician/ Assistant Professor/ Principal Investigator, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Delivery2
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Pain
Keywords: lower transverse cesarean delivery; Pregnant women
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SofPulse nonfunctional device. (Placebo Comparator): The Sofpulse non-functional device is placed over the incision after cesarean delivery and then turned on. The device only appears to be function correctly because the lights turn on, but does not emit a pulsed electromagnetic frequency..
  Interventions: Device: SofPulse
- Active (Active Comparator): The Sofpulse Pulsed electromagnetic frequency device is placed over the incision after cesarean delivery and then turned on. Device appears to be operational and functions correctly.
  Interventions: Device: SofPulse

INTERVENTIONS:
Device: SofPulse — Pulsed Electomagnetic Field Therapy Device placed over incision and turned on and kept in place with tape.

SUMMARY:
A double-blinded randomized control study using a pulsed electromagnetic field therapy to establish whether this device decreases patient pain and decreases narcotic use in women who have undergone cesarean delivery.

DETAILED DESCRIPTION:
This prospective, double-blind, randomized, sham-controlled clinical trial will investigate the effectiveness of PEMF using the Ivivi SofPulse on postoperative pain severity and narcotic use in women after cesarean delivery at Jacobi Medical Center. On admission to labor and delivery or in the obstetrical outpatient office, potential subjects will complete questions related to inclusion / exclusion criteria and sign a consent to participate in the study. If eligible, patients will receive a Ivivi Sofpulse device which will be placed over the incisional area and turned on. The devices are randomized into functional and sham groups. The device will be left around the incision site unless the patient needs to shower. In an effort to minimize bias, the patients, providers and investigators will not be aware if the device is functional or not. Lot numbers will accompany the device. After completion of the study, the Lot numbers, which will be provided by the manufacturer, will reveal which devices were functional devices or shams. These lot numbers will only be provided on completion of the trial. Wong-Baker Faces pain assessment tool will be evaluated by the Principal Investigator (PI) or co-investigator for determination of subjective postoperative pain at 0, 2, 6, 12, 24, 48, and 72 hours after cesarean delivery. Amount of oxycodone in milligrams consumed by patients will be recorded 24, 48, 72 hours after cesarean delivery. Postoperative anesthesia type (Duramorph or morphine patient controlled anesthesia pump) will be recorded as well. Subjects will be randomized to PEMF treatment (functional), or sham treatment. All subjects will be followed for the duration of their stay in the hospital following their cesarean delivery.

No follow-up is required. The goal is to recruit one hundred patients over the course of four months. Patient data will be identified by use of medical record number and will be kept private on the Jacobi Medical Center Obstetrics and Gynecology server which is password protected. Access will only be for the investigator and co-investigators in the study. Nurse on labor and delivery have already received an in-service on the proper use of this device.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years
* Female
* Undergoing lower transverse cesarean delivery or cesarean delivery with bilateral tubal ligation.
* Pfannenstiel Skin incision
* Consent to the study and willing to comply with study methods

Exclusion Criteria:

* • Subjects who have any implanted metallic leads, wires, or systems (e.g. pacemaker, implantable cardioverterdefibrillator)

  * Patients undergoing additional procedures at the time of their cesarean delivery such as cesarean hysterectomy or myomectomy.
  * Patients with vertical skin or uterine incisions.
  * Patients who forget to, or decide not to, replace PEMF device

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Pain, assessed by patients using a pain scale | 72 hours or hospital stay
  Patient uses pain scale to give subjective assesment of pain after cesarean delivery

SECONDARY OUTCOMES:
Narcotic Use | 72 hours or hospital stay
  An assesment of the amount of narcotics uses for pain control after cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Donald C Phillibert, MD, Principal Investigator — Jacobi Medical Center

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021